CLINICAL TRIAL: NCT01230697
Title: Perspective Evaluation of Hormones Involved in Serum Phosphate Homeostasis in Patients With Metastatic Renal Cells Carcinoma or Hepatocellular Carcinoma Treated With Sorafenib. Multicenter Cohort Study
Brief Title: Perspective Evaluation of Hormones Involved in Serum Phosphate Homeostasis in Patients With Metastatic Renal Cells Carcinoma or Hepatocellular Carcinoma Treated With Sorafenib (SORHORM)
Acronym: SORHORM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Alfredo Berruti, Dipartimento di Scienze Cliniche e Biologiche - Università di Torino
Other Study IDs: 662010
Record Dates: First submitted 2010-09-02; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-07

CONDITIONS: Kidney Cancer; Liver Cancer
Keywords: Advanced; hepatocarcinoma
MeSH Terms: conditions — Kidney Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum analites involved in phosphate homeostasis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sofanenib and Hypophosphatemia: Patients with advanced renal cells carcinoma and hepatocarcinoma in treatment with Sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 800mg/die oral

SUMMARY:
The study includes the recruitment of patients with advanced renal cells carcinoma and hepatocarcinoma in treatment with sorafenib. Multicenter cohort study. It is a prospective observational study.

DETAILED DESCRIPTION:
Several tyrosin kinase inhibitors are able to induce hypophosphatemia but the mechanisms underling this metabolic disorder are unknown.

Sorafenib is probably the drug in which this metabolic disturbance is most frequent. The aim of the study is identify variation of blood serum analites involved in hypophosphatemia in patients with advanced renal cells carcinoma and hepatocarcinoma in treatment with sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years
2. Histologically documented kidney cancer or hepatocarcinoma
3. Performance status more than / equal to 2
4. Life expectancy > 12 weeks
5. in patients with recent surgery, the wound should be completely healed before taking Sorafenib
6. required initial laboratory values: absolute neutrophil count > 1500/ul Platelets > 100,000/ul., Hemoglobin > 9.0 g/dl, Creatinine, SGOT, SGPT less than 2.0 X upper limit of normal Bilirubin less than/equal to upper limit of normal(ULN)
7. Appropriate patienty compliance

Exclusion Criteria:

1. myocardial infarction or significant change in anginal pattern within the last 6 months, symptomatic congestive heart failure (NYHA Class III or higher) or uncontrolled cardiac arrhythmia,
2. previous history of malignant disease with the exception of non melanoma skin cancer curatively treated,
3. significant neurologic or psychiatric diseases preventing patients to give a valid informed consent
4. Sintomatic brain metastases
5. because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded
6. patients with seizures that need medical treatment
7. History of heterologous transplantation
8. Patients with previous or active bleeding
9. Dialysis patients
10. Patients with history of primary hyperparathyroidism
11. Dysphagic patients
12. Taking more than four weeks of entry into the study of other bio-chemotherapy treatments
13. Previous treatment with Sorafenib
14. Recent (<6 months)or concomitant treatment with biphosphonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced renal cells carcinoma and hepatocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Identify the value variations of hormones involved in phosphate homeostasis during sorafenib administration | one year
  Assess the effects of sorafenib hormones involved in phosphate homeostasis

SECONDARY OUTCOMES:
Identify metabolic differences between renal cells cancer and hepatocarcinoma | one year
  identify differences in phosphate hormone behavior between renal cells cancer and hepatocarcinoma.
Identify variations on bone mass during sorafenib treatment | one year
  Assess Sorafenib effects on bone density and the relationship with phosphate related hormones
Identify correlations between phosphate related hormones and side effects during sorafenib treatment as a Measure of safety and tolerability | one year
  Identify the relationship between phpsphate hormones variation and Sorafenib side effects (e.g.asthenia, blood hypertension, skin toxicity).
Identify correlations between phosphate related hormones variations and patients outcome (TTP and overall survival) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Alfredo Berruti, Orbassano (To), Turin, Italy